CLINICAL TRIAL: NCT03299699
Title: FRATHEMO: Quality of Life and Adjustment Among Siblings of Children and Adolescents With Severe Hemophilia.
Brief Title: Quality of Life and Adjustment Among Siblings of Children and Adolescents With Severe Hemophilia
Acronym: FRATHEMO
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-06
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Severe Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe hemophilia is a rare and chronic disease characterized by spontaneous bleedings from early childhood, which may lead to various complications especially in joints. The diagnosis of this disease, but also its long term care have an impact on the relatives of the affected persons, including the siblings who bear daily the cognitive, emotional and social impacts of the disease.

Studies conducted in the framework of pediatric chronic diseases showed that siblings of affected children presented a higher prevalence of physical and psychological troubles (emotional distress, behavioral disorders, etc.) than siblings who were not concerned by a disease. Few studies have been conducted in the framework of severe hemophilia, and to our knowledge, no study addresses this issue in France.

DETAILED DESCRIPTION:
-The assessment of the quality of life would allow assessing both positive and negative impacts, by exploring in a global manner the children and adolescents functioning in various domains (physical and psychological well-being, relations with parents and friends, school…).

Regarding the specific context of hemophilia:

* Few studies have been conducted on the experience of severe hemophilia of a young patient by the siblings, and to our knowledge, no studies have been conducted in France on this topic.
* There are numerous studies concerning the impact of chronic diseases such as diabetes or cancer of a child on the siblings, contrary to those concerning rare diseases. Hemophilia, a frequent disease among rare diseases, might be an interesting model in order to understand the impact of this type of disorder on the functioning of the siblings.
* Contrary to insufficiently treated hemophilia potentially leading to disability, well-treated hemophilia might be considered as an at-risk disorder. In this specific context, the representation of the disease by the siblings might be singular.
* Parents are the major actors of the surveillance of the affected young patient in the everyday life. The transfer of parental responsibilities to healthy siblings, and its impact on the fraternal relationships might therefore be increased. Gender might have a specific modulating role on these elements (risk of transmission in female and different representation of the social role).
* Results presented in the literature are reported from studies whose representativeness of the study sample (or sample size) is questionable. The cohort of the French National Network FranceCoag represents at an international level a rare exhaustive population of persons with severe hemophilia followed over time.

Objectives The main objective of this study is to understand the mechanisms involved in the quality of the siblings' functioning and interactions in the context of severe hemophilia, in order to be able to propose adapted support modes.

The secondary (and operational) objectives are:

* To assess the impact of the functioning and interactions of the family on the quality of life (considered as a marker of the global health) reported by the siblings
* To compare the quality of life reported by siblings of children and adolescents with severe hemophilia, with the quality of life of the patients themselves, and with published reference values (age and gender-matched controls from the general population)
* To assess the emotional and social adjustment (behavioral disorders, academic success), which represents a mediator of the quality of life, among siblings
* To assess the moderating effects of gender, age, rank among siblings, time since diagnosis, quality of social support received, skills acquired to manage emotions, on quality of life as well as on the emotional and social adjustment
* To highlight clusters of siblings with different profiles of quality of life
* To propose tools, meetings and training sessions in order to support concerned families

Material and methods This study is complementary to the multicentric, observational, cross-sectional, TRANSHEMO study. TRANSHEMO focuses on the issues surrounding the transition into adulthood among young persons with severe hemophilia in France. This study also aims to identify some of the socio- cognitive, emotional, and familial determinants of a good transition into adulthood. Perceptions of older children and adolescents (aged 14-17 years old) with severe hemophilia and those of young adults (aged 20-29 years old) will be described et compared, regarding their expectations and their feelings about growing into adulthood.

The present study which is also a multicentric, observational, cross-sectional study, proposes to include the siblings [i.e. brothers, sisters, half-brothers and half-sisters (aged 8-18 years old)] of the older children and adolescents included in the TRANSHEMO study, living in the same household. The investigators will ask them to fill-up a booklet with several questionnaires, focused on quality of life. This study will allow to have preliminary results in order to extend the project to another age group of children with severe hemophilia and their siblings.

Expected results This study will allow to comprehend what the impact of the disease on the siblings could be, which is of particular interest in the global approach whose goal is to take care of and to support the affected persons and their relatives. The identification of difficulties among siblings and of their determinants will allow to detect children at risk of adjustment problem, in order to offer them an adapted support, but also to develop specific tools to support the families (brochures, meetings, therapeutic education activities).

ELIGIBILITY:
Inclusion Criteria:

* Sibling (brother, sister, half-brother or half-sister) of older children or adolescents included in the TRANSHEMO study, who lives in the same home)
* Sibling aged 8-18 years old
* Sibling affiliated to the French social security system
* Sibling whose parents are not opposed to the participation in the study

Exclusion Criteria:

* Sibling (brother, sister, half-brother or half-sister) of older children or adolescents who are not included in the TRANSHEMO study)
* Sibling aged under 8 or over 18 years old
* Sibling not affiliated to the French social security system
* Sibling whose parents are opposed to the participation in the study
* Sibling with difficulties reading and writing
* Sibling with learning disabilities

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: siblings of children and adolescents with severe hemophilia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Global quality of life | one day
  Kidscreen 10 Index, is a self-report measure, consisting of 10 items that are scored on a fivepoint scale, ranging from 1 (not at all/never) to 5 (extremely/ never)

SECONDARY OUTCOMES:
Emotional adjustment | one day
  STAI questionnaire
Coping strategies use | one day
  Kidcope checklist
Social support | one day
  Child and Adolescent Social Support Scale

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France